CLINICAL TRIAL: NCT01067781
Title: A Phase 2, Gender-Stratified, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Immunogenicity of a Two Vaccination Regimen With the Travelers' Diarrhea Vaccine System in Healthy Adults
Brief Title: Safety and Immunogenicity Study of Traveler's Diarrhea Vaccine Patch
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intercell USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ELT208
Record Dates: First submitted 2010-02-09; First posted 2010-02-12 (Estimated); Results first posted 2014-03-13 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Diarrhea
Keywords: Prevention of Travelers' Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Two vaccination regimen with an LT patch (no swabbing)
  Interventions: Biological: Heat-Labile Enterotoxin of E. coli (LT)
- 2 (Experimental): Two vaccination regimen with an LT patch (with swabbing)
  Interventions: Biological: Heat-Labile Enterotoxin of E. coli (LT)
- 3 (Placebo Comparator): Two vaccination regimen with a placebo patch (no swabbing)
  Interventions: Biological: Placebo
- 4 (Placebo Comparator): Two vaccination regimen with a placebo patch (with swabbing)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Heat-Labile Enterotoxin of E. coli (LT) — Travelers' Diarrhea Vaccine System
  Arms: 1; 2
Biological: Placebo — Travelers' Diarrhea Vaccine System
  Arms: 3; 4

SUMMARY:
The purpose of this study is to evaluate and compare the safety and immune responses following a two vaccination regimen by transcutaneous immunization with heat-labile enterotoxin of E. coli (LT) patches or Placebo, with or without alcohol swabbing

ELIGIBILITY:
Inclusion Criteria:

1. A female or male 18-64 (inclusive) years of age;
2. In good health as determined by medical history and screening exam;
3. Females who are post-menopausal, surgically sterile, or have a negative serum/urine pregnancy test at Day 0 and agree not to become pregnant for the duration of study.

Exclusion Criteria:

1. Abnormalities at physical exam [as determined by the Toxicity Grading Scale (Grade 1-4)];
2. Laboratory abnormalities [as determined by the Toxicity Grading Scale (Grade 1 4)] at screening;
3. Participated in research involving investigational product within 30 days before planned date of first vaccination;
4. Ever received investigational enterotoxigenic E. coli, LT, or LT (R192G) or NasalFlu, Berna Biotech, Ltd;
5. Women who are pregnant or breastfeeding;
6. Clinically significant underlying enteric, pulmonary, cardiac or renal disease;
7. Current seizure disorder;
8. Current use of immunosuppressive therapy (inhaled steroids are allowed);
9. Known or suspected alcohol abuse or illicit drug use within the last year;
10. Positive Serology for HIV-1, HIV-2, HbsAg, or HCV;
11. Known allergies to any component of the vaccine including adhesives;
12. An employee of the study site;
13. An employee of Intercell (global) or an immediate family member;
14. Visible tattoos or marks (tattoos/scars) at the vaccination areas that would prevent appropriate dermatologic monitoring of the vaccination sites;
15. Receipt of any routine vaccinations within 7 days prior to, or following, the date of planned study vaccinations.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2010-02; Primary Completion 2010-09 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sheldon, MD, Principal Investigator — Miami Research Associates
Locations (5):
- United States (5):
  - Advanced Clinical Research Institute, Anaheim, California
  - Miami Research Associates, South Miami, Florida
  - Johnson County Clinical Trials, Lenexa, Kansas
  - Radiant Research, Cincinnati, Ohio
  - Clinical Trials of Texas, San Antonio, Texas

REFERENCES:
- See also: Intercell Home Page — http://www.valneva.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: 37.5μg LT, No Swab: Two vaccination regimen with an LT patch (no swabbing)
  Heat-Labile Enterotoxin of E. coli (LT): Travelers' Diarrhea Vaccine System
- Group 2: 37.5μg LT, Swab: Two vaccination regimen with an LT patch (with swabbing)
  Heat-Labile Enterotoxin of E. coli (LT): Travelers' Diarrhea Vaccine System
- Group 3: 0μg LT, No Swab: Two vaccination regimen with a placebo patch (no swabbing)
  Placebo: Travelers' Diarrhea Vaccine System
- Group 4: 0μg LT, Swab: Two vaccination regimen with a placebo patch (with swabbing)
  Placebo: Travelers' Diarrhea Vaccine System
Period: Up to Day 180
Arm/Group | Group 1: 37.5μg LT, No Swab | Group 2: 37.5μg LT, Swab | Group 3: 0μg LT, No Swab | Group 4: 0μg LT, Swab
Started | 203 | 199 | 97 | 101
Completed | 173 | 168 | 89 | 89
Not Completed | 30 | 31 | 8 | 12
Period: 180 to Day 720
Arm/Group | Group 1: 37.5μg LT, No Swab | Group 2: 37.5μg LT, Swab | Group 3: 0μg LT, No Swab | Group 4: 0μg LT, Swab
Started | 173 | 168 | 89 | 89
Completed | 3 (all subjects followed till Day180;if ongoing local AE, FU every 6 mths till AE resolved (max.Day720)) | 4 (all subjects followed till Day180;if ongoing local AE, FU every 6 mths till AE resolved (max.Day720)) | 0 (all subjects followed till Day180;if ongoing local AE, FU every 6 mths till AE resolved (max.Day720)) | 0 (all subjects followed till Day180;if ongoing local AE, FU every 6 mths till AE resolved (max.Day720))
Not Completed | 170 | 164 | 89 | 89

BASELINE CHARACTERISTICS:
Population: safety population: includes all study subjects that were consented and received investigational study material (i.e., at least one vaccination)
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 37.5μg LT, No Swab | Group 2: 37.5μg LT, Swab | Group 3: 0μg LT, No Swab | Group 4: 0μg LT, Swab | Total
Number analyzed (Participants) | 203 | 199 | 97 | 101 | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (12.8) | 35.3 (13.1) | 35.0 (13.6) | 35.7 (12.8) | 35.3 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 99 | 48 | 51 | 300
  Male | 101 | 100 | 49 | 50 | 300

OUTCOME MEASURES:

1. Primary Outcome: Characterization and Comparison of the Safety of the TD Vaccine System: (1) Solicited and Unsolicited Adverse Events (AEs) (2) Clinical Laboratory Safety (3) Serious AEs
Description: Erythema, rash, pain, pruritus, hyperpigmentation, hypopigmentation and edema were solicited local AEs for the duration of the study. Fever, malaise, headache, and diarrhea were solicited systemic AEs for the first seven days following each vaccination; events reported outside this time frame were considered non-solicited.
Time Frame: Day 0 to Day 180
Measure: Number; unit: participants
Groups:
- Group 1 & 2 Combined: 37.5µg LT Patch; Group 3 & 4 Combined: Placebo Patch (0µg LT): with or without swabbing
Arm/Group | Group 1 & 2 Combined: 37.5µg LT Patch | Group 3 & 4 Combined: Placebo Patch (0µg LT)
Number analyzed (Participants) | 402 | 198
participants
  Solicited Local Adverse Events (1st vaccination) | 318 | 93
  Solicited Local AEs (2nd vaccination) | 327 | 62
  Non-solicited Local AEs (1st vaccination) | 20 | 3
  Non-solicited Local AEs (2nd vaccination) | 11 | 3
  Solicited Systemic AEs (overall) | 134 | 59
  Non-solicited Systemic AEs (overall) | 296 | 148
  Serious AEs | 4 | 0

2. Secondary Outcome: Characterization and Comparison of Group LT-specific Immune Responses to the TD Vaccine System: Geometric Mean Titers
Description: LT immunoglobulin G (IgG) and immunoglobulin A (IgA)
Time Frame: Day 0 to Day 180
Population: the numbers analyzed differs from the Overall number analyzed because for this the Immunogenicity Evaluable Population (IEP) was used: includes all study subjects that were consented, randomized, received the assigned Treatments (both vaccinations) without significant protocol deviations and had blood drawn on Day 0, Day 21 and Day 35
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- LT Patch Without Swabbing: Two vaccination (Day 0 and Day 14) regimen with an LT patch (no swabbing), 37.5 mcg LT
  Heat-Labile Enterotoxin of E. coli (LT): Travelers' Diarrhea Vaccine System
- LT Patch With Swabbing: Two vaccination (Day 0 and Day 14) regimen with an LT patch (with swabbing), 37.5 mcg LT
  SPS:Buffer-prepared site swabbed with a 70% isopropyl alcohol pad
  Heat-Labile Enterotoxin of E. coli (LT): Travelers' Diarrhea Vaccine System
- Placebo Patch Without Swabbing: Two vaccination (Day 0 and Day 14) regimen with a placebo patch (no swabbing)
  Placebo: Travelers' Diarrhea Vaccine System
- Placebo Patch With Swabbing: Two vaccination (Day 0 and Day 14) regimen with a placebo patch (with swabbing)
  SPS:Buffer-prepared site swabbed with a 70% isopropyl alcohol pad
  Placebo: Travelers' Diarrhea Vaccine System
Arm/Group | LT Patch Without Swabbing | LT Patch With Swabbing | Placebo Patch Without Swabbing | Placebo Patch With Swabbing
Number analyzed (Participants) | 182 | 173 | 92 | 90
titers
  IgG Day 0 | 442.21 [386.83 to 505.53] | 421.20 [368.78 to 481.06] | 435.64 [360.89 to 525.89] | 344.40 [282.43 to 419.98]
  IgG Day 7: number analyzed (Participants) | 181 | 172 | 90 | 89
  IgG Day 7 | 455.68 [402.07 to 516.44] | 437.80 [380.75 to 503.39] | 426.28 [352.98 to 514.81] | 348.13 [289.47 to 418.67]
  IgG Day 14: number analyzed (Participants) | 181 | 172 | 92 | 90
  IgG Day 14 | 1042.41 [862.90 to 1259.26] | 1148.98 [940.12 to 1404.24] | 433.13 [357.98 to 524.06] | 336.41 [276.48 to 409.34]
  IgG Day 21 | 2036.77 [1678.75 to 2471.14] | 2537.89 [2073.46 to 3106.35] | 447.47 [371.36 to 539.18] | 404.66 [332.68 to 492.21]
  IgG Day 28: number analyzed (Participants) | 180 | 172 | 92 | 90
  IgG Day 28 | 4010.55 [3424.12 to 4697.41] | 4806.53 [4057.60 to 5693.69] | 571.09 [463.60 to 703.49] | 418.78 [353.08 to 496.69]
  IgG Day 35 | 4820.85 [4121.82 to 5638.42] | 6005.34 [5126.11 to 7035.37] | 573.03 [471.04 to 697.12] | 421.34 [359.37 to 494.01]
  IgG Day 42: number analyzed (Participants) | 181 | 170 | 90 | 90
  IgG Day 42 | 5229.02 [4526.96 to 6039.96] | 5757.21 [4949.95 to 6696.11] | 582.72 [469.17 to 723.76] | 427.64 [357.27 to 511.86]
  IgG Day 56: number analyzed (Participants) | 177 | 167 | 90 | 90
  IgG Day 56 | 5056.13 [4380.77 to 5835.60] | 5633.07 [4910.89 to 6461.46] | 588.69 [484.87 to 714.74] | 411.26 [340.90 to 496.15]
  IgG Day 90: number analyzed (Participants) | 169 | 161 | 89 | 89
  IgG Day 90 | 4833.84 [4231.66 to 5521.71] | 4695.02 [4085.96 to 5394.87] | 537.23 [440.47 to 655.24] | 464.11 [390.50 to 551.61]
  IgG Day 180: number analyzed (Participants) | 161 | 154 | 85 | 86
  IgG Day 180 | 2809.18 [2440.40 to 3233.67] | 2843.59 [2486.76 to 3251.61] | 498.20 [404.73 to 613.24] | 419.89 [354.80 to 496.93]
  IgA Day 0 | 72.71 [65.10 to 81.22] | 67.06 [60.62 to 74.18] | 63.00 [55.53 to 71.46] | 69.52 [59.90 to 80.69]
  IgA Day 7: number analyzed (Participants) | 181 | 172 | 90 | 89
  IgA Day 7 | 74.30 [66.09 to 83.52] | 65.29 [58.70 to 72.62] | 62.26 [54.81 to 70.72] | 70.77 [60.62 to 82.61]
  IgA Day 14: number analyzed (Participants) | 181 | 172 | 92 | 90
  IgA Day 14 | 130.89 [112.10 to 152.83] | 132.33 [111.62 to 156.87] | 59.70 [53.47 to 66.67] | 69.79 [59.78 to 81.48]
  IgA Day 21 | 183.42 [155.55 to 216.29] | 175.05 [147.46 to 207.79] | 65.82 [56.12 to 77.18] | 69.91 [59.83 to 81.68]
  IgA Day 28: number analyzed (Participants) | 180 | 172 | 92 | 90
  IgA Day 28 | 290.95 [251.96 to 335.99] | 294.68 [252.19 to 344.34] | 67.52 [57.86 to 78.79] | 76.00 [64.41 to 89.66]
  IgA Day 35 | 284.26 [247.37 to 326.66] | 286.88 [245.46 to 335.29] | 69.84 [60.23 to 80.99] | 74.91 [63.19 to 88.81]
  IgA Day 42: number analyzed (Participants) | 181 | 170 | 90 | 90
  IgA Day 42 | 248.33 [214.74 to 287.17] | 261.53 [223.84 to 305.58] | 67.45 [58.30 to 78.03] | 71.97 [61.24 to 84.57]
  IgA Day 56: number analyzed (Participants) | 177 | 167 | 90 | 90
  IgA Day 56 | 229.76 [198.94 to 265.34] | 232.70 [200.49 to 270.09] | 70.11 [59.62 to 82.44] | 78.60 [66.30 to 93.20]
  IgA Day 90: number analyzed (Participants) | 169 | 161 | 89 | 89
  IgA Day 90 | 168.18 [144.93 to 195.16] | 166.85 [142.94 to 194.75] | 61.79 [53.98 to 70.73] | 70.93 [60.92 to 82.59]
  IgA Day 180: number analyzed (Participants) | 161 | 154 | 85 | 86
  IgA Day 180 | 120.12 [104.49 to 138.08] | 124.50 [107.41 to 144.30] | 56.00 [50.00 to 62.72] | 61.30 [53.98 to 69.60]

3. Secondary Outcome: Characterization and Comparison of Group LT-specific Immune Responses to the TD Vaccine System: Geometric Mean Fold Ratios
Description: LT immunoglobulin G (IgG) and immunoglobulin A (IgA)
Time Frame: Day 0 to Day 180
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Fold Ratios (GMFRs)
Arm/Group | LT Patch Without Swabbing | LT Patch With Swabbing | Placebo Patch Without Swabbing | Placebo Patch With Swabbing
Number analyzed (Participants) | 182 | 173 | 92 | 90
Geometric Mean Fold Ratios (GMFRs)
  LT IgG Day 7: number analyzed (Participants) | 181 | 172 | 90 | 89
  LT IgG Day 7 | 1.02 [0.95 to 1.09] | 1.04 [0.97 to 1.12] | 0.96 [0.89 to 1.04] | 1.02 [0.95 to 1.10]
  LT IgG Day 14: number analyzed (Participants) | 181 | 172 | 92 | 90
  LT IgG Day 14 | 2.37 [2.01 to 2.81] | 2.73 [2.26 to 3.31] | 0.99 [0.92 to 1.07] | 0.98 [0.90 to 1.06]
  LT IgG Day 21 | 4.61 [3.76 to 5.65] | 6.03 [4.86 to 7.47] | 1.03 [0.94 to 1.12] | 1.17 [1.05 to 1.32]
  LT IgG Day 28: number analyzed (Participants) | 180 | 172 | 92 | 90
  LT IgG Day 28 | 8.91 [7.35 to 10.81] | 11.39 [9.33 to 13.9] | 1.31 [1.08 to 1.58] | 1.22 [1.08 to 1.37]
  LT IgG Day 35 | 10.90 [8.94 to 13.29] | 14.26 [11.74 to 17.31] | 1.32 [1.13 to 1.53] | 1.22 [1.08 to 1.38]
  LT IgG Day 42: number analyzed (Participants) | 181 | 170 | 90 | 90
  LT IgG Day 42 | 11.72 [9.67 to 14.21] | 13.65 [11.33 to 16.44] | 1.36 [1.11 to 1.66] | 1.24 [1.09 to 1.41]
  LT IgG Day 56: number analyzed (Participants) | 177 | 167 | 90 | 90
  LT IgG Day 56 | 11.34 [9.40 to 13.68] | 13.47 [11.26 to 16.10] | 1.36 [1.15 to 1.60] | 1.19 [1.05 to 1.36]
  LT IgG Day 90: number analyzed (Participants) | 169 | 161 | 89 | 89
  LT IgG Day 90 | 11.18 [9.38 to 13.32] | 11.04 [9.28 to 13.15] | 1.23 [1.12 to 1.36] | 1.36 [1.20 to 1.54]
  LT IgG Day 180: number analyzed (Participants) | 161 | 154 | 85 | 86
  LT IgG Day 180 | 6.49 [5.41 to 7.79] | 6.58 [5.58 to 7.76] | 1.15 [1.01 to 1.30] | 1.23 [1.09 to 1.40]
  LT IgA Day 7: number analyzed (Participants) | 181 | 172 | 90 | 89
  LT IgA Day 7 | 1.02 [0.96 to 1.08] | 0.98 [0.93 to 1.04] | 1.00 [0.93 to 1.06] | 1.02 [0.97 to 1.08]
  LT IgA Day 14: number analyzed (Participants) | 181 | 172 | 92 | 90
  LT IgA Day 14 | 1.81 [1.59 to 2.07] | 1.99 [1.69 to 2.34] | 0.95 [0.88 to 1.02] | 1.00 [0.94 to 1.07]
  LT IgA Day 21 | 2.52 [2.17 to 2.93] | 2.61 [2.20 to 3.10] | 1.04 [0.92 to 1.19] | 1.01 [0.93 to 1.08]
  LT IgA Day 28: number analyzed (Participants) | 180 | 172 | 92 | 90
  LT IgA Day 28 | 4.03 [3.49 to 4.65] | 4.38 [3.72 to 5.17] | 1.07 [0.96 to 1.20] | 1.09 [1.00 to 1.20]
  LT IgA Day 35 | 3.91 [3.41 to 4.48] | 4.28 [3.63 to 5.04] | 1.11 [0.99 to 1.24] | 1.08 [0.98 to 1.18]
  LT IgA Day 42: number analyzed (Participants) | 181 | 170 | 90 | 90
  LT IgA Day 42 | 3.41 [2.96 to 3.92] | 3.92 [3.34 to 4.61] | 1.07 [0.97 to 1.19] | 1.04 [0.93 to 1.15]
  LT IgA Day 56: number analyzed (Participants) | 177 | 167 | 90 | 90
  LT IgA Day 56 | 3.16 [2.76 to 3.62] | 3.53 [3.03 to 4.11] | 1.13 [1.01 to 1.27] | 1.13 [1.01 to 1.27]
  LT IgA Day 90: number analyzed (Participants) | 169 | 161 | 89 | 89
  LT IgA Day 90 | 2.32 [2.03 to 2.65] | 2.58 [2.22 to 3.0] | 0.98 [0.92 to 1.06] | 1.02 [0.92 to 1.12]
  LT IgA Day 180: number analyzed (Participants) | 161 | 154 | 85 | 86
  LT IgA Day 180 | 1.66 [1.46 to 1.89] | 1.89 [1.65 to 2.16] | 0.92 [0.83 to 1.03] | 0.90 [0.80 to 1.00]

4. Secondary Outcome: Characterization and Comparison of Group LT-specific Immune Responses to the TD Vaccine System: Seroconversion Rates
Description: LT immunoglobulin G (IgG) and immunoglobulin A (IgA)
Time Frame: Day 0 to Day 180
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | LT Patch Without Swabbing | LT Patch With Swabbing | Placebo Patch Without Swabbing | Placebo Patch With Swabbing
Number analyzed (Participants) | 182 | 173 | 92 | 90
percentage of participants
  LT IgG Day 7: number analyzed (Participants) | 181 | 172 | 90 | 89
  LT IgG Day 7 | 7.18 [3.88 to 11.97] | 7.56 [4.09 to 12.58] | 3.33 [0.69 to 9.43] | 6.74 [2.51 to 14.10]
  LT IgG Day 14: number analyzed (Participants) | 181 | 172 | 92 | 90
  LT IgG Day 14 | 47.51 [40.06 to 55.05] | 49.42 [41.72 to 57.13] | 2.17 [0.26 to 7.63] | 3.33 [0.69 to 9.43]
  LT IgG Day 21 | 67.03 [59.69 to 73.81] | 74.57 [67.40 to 80.87] | 5.43 [1.79 to 12.23] | 16.67 [9.64 to 26.00]
  LT IgG Day 28: number analyzed (Participants) | 180 | 172 | 92 | 90
  LT IgG Day 28 | 86.67 [80.81 to 91.27] | 89.53 [83.97 to 93.68] | 14.13 [7.74 to 22.95] | 16.67 [9.64 to 26.00]
  LT IgG Day 35 | 90.11 [84.82 to 94.03] | 93.06 [88.20 to 96.36] | 15.22 [8.58 to 24.21] | 17.78 [10.52 to 27.26]
  LT IgG Day 42: number analyzed (Participants) | 181 | 170 | 90 | 90
  LT IgG Day 42 | 90.61 [85.39 to 94.43] | 94.71 [90.19 to 97.55] | 17.78 [10.52 to 27.26] | 20.00 [12.31 to 29.75]
  LT IgG Day 56: number analyzed (Participants) | 177 | 167 | 90 | 90
  LT IgG Day 56 | 92.09 [87.09 to 95.61] | 95.81 [91.55 to 98.30] | 16.67 [9.64 to 26.00] | 16.67 [9.64 to 26.00]
  LT IgG Day 90: number analyzed (Participants) | 169 | 161 | 89 | 89
  LT IgG Day 90 | 93.49 [88.65 to 96.71] | 93.79 [88.87 to 96.98] | 11.24 [5.52 to 19.69] | 24.72 [16.19 to 35.00]
  LT IgG Day 180: number analyzed (Participants) | 161 | 154 | 85 | 86
  LT IgG Day 180 | 85.09 [78.64 to 90.21] | 90.26 [84.44 to 94.45] | 9.41 [4.15 to 17.71] | 20.93 [12.90 to 31.05]
  LT IgA Day 7: number analyzed (Participants) | 181 | 172 | 90 | 89
  LT IgA Day 7 | 1.66 [0.34 to 4.77] | 1.74 [0.36 to 5.01] | 0.00 [0.00 to 4.02] | 0.00 [0.00 to 4.06]
  LT IgA Day 14: number analyzed (Participants) | 181 | 172 | 92 | 90
  LT IgA Day 14 | 17.68 [12.42 to 24.03] | 23.84 [17.68 to 30.92] | 0.00 [0.00 to 3.93] | 1.11 [0.03 to 6.04]
  LT IgA Day 21 | 32.42 [25.68 to 39.74] | 36.42 [29.25 to 44.06] | 1.09 [0.03 to 5.91] | 1.11 [0.03 to 6.04]
  LT IgA Day 28: number analyzed (Participants) | 180 | 172 | 92 | 90
  LT IgA Day 28 | 50.56 [43.02 to 58.07] | 54.65 [46.90 to 62.24] | 2.17 [0.26 to 7.63] | 2.22 [0.27 to 7.80]
  LT IgA Day 35 | 51.10 [43.60 to 58.57] | 54.91 [47.18 to 62.48] | 2.17 [0.26 to 7.63] | 2.22 [0.27 to 7.80]
  LT IgA Day 42: number analyzed (Participants) | 181 | 170 | 90 | 90
  LT IgA Day 42 | 46.96 [39.52 to 54.51] | 51.76 [43.99 to 59.48] | 1.11 [0.03 to 6.04] | 2.22 [0.27 to 7.80]
  LT IgA Day 56: number analyzed (Participants) | 177 | 167 | 90 | 90
  LT IgA Day 56 | 40.68 [33.37 to 48.30] | 49.70 [41.88 to 57.53] | 3.33 [0.69 to 9.43] | 3.33 [0.69 to 9.43]
  LT IgA Day 90: number analyzed (Participants) | 169 | 161 | 89 | 89
  LT IgA Day 90 | 26.63 [20.13 to 33.96] | 37.27 [29.79 to 45.23] | 0.00 [0.00 to 4.06] | 1.12 [0.03 to 6.10]
  LT IgA Day 180: number analyzed (Participants) | 161 | 154 | 85 | 86
  LT IgA Day 180 | 14.91 [9.79 to 21.36] | 17.53 [11.88 to 24.47] | 1.18 [0.03 to 6.38] | 0.00 [0.00 to 4.20]

ADVERSE EVENTS:
Arm/Group | Group 1: 37.5μg LT, No Swab | Group 2: 37.5μg LT, Swab | Group 3: 0μg LT, No Swab | Group 4: 0μg LT, Swab
Serious Adverse Events (participants affected / at risk) | 1/203 | 3/199 | 0/97 | 0/101
Other Adverse Events (participants affected / at risk) | 197/203 | 192/199 | 90/97 | 92/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 37.5μg LT, No Swab (N=203) | Group 2: 37.5μg LT, Swab (N=199) | Group 3: 0μg LT, No Swab (N=97) | Group 4: 0μg LT, Swab (N=101)
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Accelerated hypertension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: 37.5μg LT, No Swab (N=203) | Group 2: 37.5μg LT, Swab (N=199) | Group 3: 0μg LT, No Swab (N=97) | Group 4: 0μg LT, Swab (N=101)
Headache (Nervous system disorders) | 33 | 36 | 19 | 18
Malaise (General disorders) | 18 | 25 | 9 | 6
Diarrhea (Gastrointestinal disorders) | 33 | 40 | 14 | 14
Vaccination site erythema (General disorders) | 164 | 157 | 44 | 32
Vaccination site rash (General disorders) | 173 | 168 | 9 | 10
Vaccination site hyperpigmentation (General disorders) | 139 | 138 | 6 | 6
Vaccination site edema (General disorders) | 56 | 73 | 2 | 1
Vaccination site pain (General disorders) | 40 | 47 | 10 | 13
Vaccination site pruritis (General disorders) | 163 | 156 | 22 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other